CLINICAL TRIAL: NCT03040713
Title: 18F-AV-1451 PET Imaging in Subjects With Frontotemporal Dementia
Brief Title: Flortaucipir PET Imaging in Subjects With FTD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A19
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FTD Subjects (Experimental): Subjects diagnosed by dementia specialist with a clinical Frontotemporal Dementia (FTD) syndrome and expected tau or tar DNA binding protein (TDP)-43 pathology receiving a flortaucipir PET scan
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq)(10 millicurie [mCi]) injection, single dose
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This study is designed to assess the usefulness of flortaucipir in Positron Emission Tomography (PET) imaging for subjects diagnosed with Frontotemporal Dementia (FTD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed by a dementia specialist with symptomatic clinical syndromes with expected Frontotemporal Dementia (FTD) pathology will be enrolled. Clinical syndromes associated with FTD pathology include: behavioral-variant FTD, FTD with motor-neuron disease, non-fluent/agrammatic and semantic variants of primary progressive aphasia, progressive supranuclear palsy syndrome and corticobasal syndrome.
* Have provided informed consent or have a legally authorized (LAR) provide consent for study procedures
* Have had volumetric brain MRI obtained in site's companion protocol within one year of enrollment
* Can tolerate PET scan procedures

Exclusion Criteria:

* Have clinically significant cardiac, hepatic, renal, pulmonary, metabolic, or endocrine disturbances that pose potential safety risk
* Have history of risk factors for Torsades de Pointes (TdP) or taking medication known to cause QT prolongation
* Have history of drug or alcohol dependence within the last year
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using reliable contraception
* Have history of relevant severe drug allergy or hypersensitivity
* Have received an investigational medication under FDA IND protocol within 30 days of planned imaging session
* Have received a radiopharmaceutical for imaging/therapy within 24 hours of imaging session
* Possess PET scan evidence of amyloid deposition
* Determined by the investigator to be unsuitable for this type of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Movement Disorder Center, UCSD, La Jolla, California
  - Memory and Aging Center, UCSF, San Francisco, California
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Soleimani-Meigooni DN, Iaccarino L, La Joie R, Baker S, Bourakova V, Boxer AL, Edwards L, Eser R, Gorno-Tempini ML, Jagust WJ, Janabi M, Kramer JH, Lesman-Segev OH, Mellinger T, Miller BL, Pham J, Rosen HJ, Spina S, Seeley WW, Strom A, Grinberg LT, Rabinovici GD. 18F-flortaucipir PET to autopsy comparisons in Alzheimer's disease and other neurodegenerative diseases. Brain. 2020 Dec 5;143(11):3477-3494. doi: 10.1093/brain/awaa276. PMID 33141172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Apr 2017 and Oct 2018.
Pre-assignment Details: As a result of a positive amyloid scan at screening, 1 subject was discontinued prior to administration of flortaucipir. Two additional subjects had positive amyloid scans and received flortaucipir, but were excluded from the per protocol population results (n=13).
Period: Overall Study
Arm/Group | FTD Subjects
Started | 16
Completed | 13
Not Completed | 3
Not completed — Positive amyloid scan | 3

BASELINE CHARACTERISTICS:
Population: All subjects receiving one dose of flortaucipir in the study
Groups:
- FTD Subjects: Subjects diagnosed by dementia specialist with a clinical Frontotemporal Dementia (FTD) syndrome and expected tau or TDP-43 pathology receiving a flortaucipir PET scan
Arm/Group | FTD Subjects
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 25.6 (6.38)

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Evaluation of Flortaucipir PET Scans
Description: Subject scans were visually evaluated by an expert reader into three groups. Advanced Alzheimer's Disease (AD) scan pattern = In either hemisphere, increased neocortical activity in the parietal/precuneus region(s), or frontal region(s) with increased uptake in the posterolateral temporal (PLT), parietal, or occipital region(s). Moderate AD scan pattern = In either hemisphere, increased neocortical activity limited to the PLT or occipital region(s). Not AD scan pattern = No increased neocortical activity, or increased neocortical activity isolated to the mesial temporal, anterolateral temporal, and/or frontal regions.
Time Frame: baseline scan
Measure: Count of Participants; unit: Participants
Arm/Group | FTD Subjects
Number analyzed (Participants) | 13
Participants
  Advanced AD Scan Pattern (τAD++) | 0
  Moderate AD Scan Pattern (τAD+) | 0
  Not AD Scan Pattern (τAD-) | 13

2. Primary Outcome: Quantitative Evaluation of Flortaucipir PET Scans
Description: Standard Uptake Value Ratio (SUVr) using a weighted cortical average (MUBADA), and individual regions. For SUVr, a value of 1 or lower signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan
Population: All amyloid negative FTD subjects who had a PET scan that was able to be quantitatively evaluated (n=12). One subject did not have magnetic resonance imaging available, so quantitation was not possible.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | FTD Subjects
Number analyzed (Participants) | 12
standardized uptake value ratio (SUVr)
  MUBADA | 1.00903 (0.036582)
  Parietal | 0.91992 (0.054753)
  Temporal | 0.94920 (0.041189)
  Frontal | 0.89825 (0.086118)
  Caudate | 0.63508 (0.130466)

ADVERSE EVENTS:
Time Frame: AEs were collected at scan visit and for 48 hours after flortaucipir administration.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection, at an imaging visit. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- FTD Subjects Safety Population: Subjects diagnosed with a clinical Frontotemporal Dementia (FTD) syndrome and expected tau or TDP-43 pathology receiving a flortaucipir PET scan
Arm/Group | FTD Subjects Safety Population
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTD Subjects Safety Population (N=15)
Feeling cold (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT03040713/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT03040713/SAP_001.pdf